CLINICAL TRIAL: NCT04859348
Title: Effects of Antenatal Exercises on Clinical Outcomes in Pregnant Females With Gestational Diabetes Mellitus: a Randomized Controlled Trial
Brief Title: Effects of Antenatal Exercises on Clinical Outcomes in Pregnant Females With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/600-1/2020
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Gestational Diabetes
Keywords: Antenatal Exercise; APGAR Score; C-section; Mode of delivery; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: G- A 36 participants received only routine treatment for GDM G- B 36 participants receive routine therapy (insulin therapy and diet control) and Aerobic and strengthening Exercises.
Who Masked: Outcomes Assessor
Masking Description: outcomes accessor donot know the type of intervention given to patient not during evaluation or data record
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A ( RPT+ Insulin Therapy) (Experimental): Group A includes participants received the routine physical therapy only.
  Interventions: Other: routine physical therapy
- Group-B (RPT+ Antenatal Exercises+ Insulin therapy) (Experimental): Group B includes participants were given antenatal exercise program from 20- 24 weeks of gestation to till the date of delivery, with addition of the routine physical therapy plan.
  Interventions: Other: routine physical therapy and antenatal exercises

INTERVENTIONS:
Other: routine physical therapy — G- A 36 participants received only routine treatment for GDM which includes insulin therapy and diet control guided by gynecologist and routine physical therapy which includes walk for 1 hr with proper warm up and cool down periods, three times in a week from 20-24 weeks of gestation to till delivery.
  Arms: Group-A ( RPT+ Insulin Therapy)
Other: routine physical therapy and antenatal exercises — G- B 36 participants receive routine therapy (insulin therapy and diet control) and Aerobic and strengthening Exercises for 3 days a week, for 2 weeks 6 sessions under the supervision of physiotherapist and remaining was performed at home. Exercise was started from 15 min and reach to 30 mins gradually.10-15-minute warm-up, cool-down period was included by using ACOG Guideline. Aerobic exercise includes a brisk walk and strengthening exercise were performed with hold for 5 seconds and 10 repetitions. Exercise should stop if they experience any signs of dizziness, dyspnea, amniotic fluid leaking or vaginal bleeding. Confidentiality and blindness ensure by random allocation.
  Arms: Group-B (RPT+ Antenatal Exercises+ Insulin therapy)

SUMMARY:
Gestational diabetes mellitus (GDM) GDM is the most common complication that affects the health of the child and mother during pregnancy. Objectives was to determine the effects of Antenatal exercises on glucose levels, mode of delivery and APGAR Score in females with gestational diabetes mellitus.

This Randomized controlled trial study was conducted on N= 72 pregnant females at department of Gynecology and Obstetrics, Mian Munshi DHQ Hospital, Lahore after Ethical approval of synopsis from institutional Review Board of the University of Lahore . The data was entered and analyzed using SPSS Version 24. .

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as glucose intolerance resulting in hyperglycemia of variable severity with onset during pregnancy. During pregnancy, GDM is the most common complication occurs and it affects the health of the child and mother.

This study aim was to investigate the effect of antenatal exercise on clinical outcomes in pregnant females with gestational diabetes mellitus.

Study Design: Randomized controlled trial. Settings: It was conducted at department of Gynecology and Obstetrics, Mian Munshi DHQ Hospital, Lahore.

Sample Size:

The calculated sample size is 30 in each group using APGAR scale as outcome measure. After adding 20% drop out the sample size will become 30+6 = 36 in each group.

Sampling Technique: Purposive sampling technique

Outcome measuring Tools -

• APGAR scale DATA COLLECTION PROCEDURE

All the participants visited from the gynecology department after the diagnosis of GDM was considered after the initial screening test. Following the inclusion and exclusion criteria before adding them to the study. These patients were allotted in two groups i.e. group A and group B via the lottery method. Informed consent were taken in written form showing that they are willing to participate in the study. The therapist had assessed the patients before the start of rehabilitation program:

Group A includes participants received the routine physical therapy only. Group B includes participants were given exercise program from 20- 24 weeks of gestation to till the date of delivery, with addition of the routine physical therapy plan.

Group A: Routine Physical Therapy (RPT) + Insulin therapy Group A- (n=36) participants received only routine treatment for gestational diabetes mellitus which includes insulin therapy and diet control programs guided by a gynecologist and routine physical therapy which includes walk for 1 hr which includes proper warm up and cool down periods, three times in a week from 20-24 weeks of gestation to till delivery.

Group -B-Antenatal + RPT + Insulin therapy+ Exercise Group B- (n=36) participants completed routine therapy and antenatal exercises which includes Aerobic and strengthening Exercises with workout 3 days a week, for 2 weeks (6 sessions under the supervision of physiotherapist and remaining was performed at home along with routine treatment for gestational diabetes mellitus which includes insulin therapy and diet control program as guided by gynecologist. The exercise program was started with quarter-hour moderate-intensity aerobic activity and slowly rising the duration to a maximum of half-hour each exercise session. A 10-15-minute warm-up physical exercise, and a 10-15-minute cool-down period was included. The duration of the exercise was assessed by using target pulse rate, the Borg scale (rate of perceived exertion), or the 'talk test.' American College of Obstetricians and Gynecologists Guideline corresponded to exercise of moderate-intensity were followed. Aerobic exercise includes a brisk walk to train the main muscle groups which includes, chest muscles, deltoid, quadriceps, and calf muscles were targeted the main muscle groups .In sitting position, strengthening exercise were performed in which one end of the Thera band was placed under the foot, hold for 5 seconds then released along with 10 repetitions. The movements were involvement of wall push-ups, shoulder flexion, shoulder abduction, knee extension and ankle plantar flexion. It was guided that pregnant women avoid exercise promptly if they experience any signs such as dizziness, dyspnea, amniotic fluid leaking or vaginal bleeding. Besides, group participant will wear loose-fitting clothing and keep hydrated while exercising in an environment with adequate temperature and moisture. All sessions of the exercise under supervision were fully documented on successful completion.

Confidentiality of all the details were ensured. A blind study (to remove chance of bias), in which random allocation of women between two categories, via the lottery system was executed.

Follow Ups Total 3 sessions per week were given to the patients for 60 min., from 20- 24 weeks of gestation to till the time of delivery. Home plan was given to the participants and follow up was done whenever participants came to gynecology department.

PROFORMA/QUESTIONNAIRE

Title "Effects of Antenatal exercises on clinical outcomes in pregnant females with gestational diabetes mellitus: A Randomized Controlled Trial" Name………………... Age …………………. Height ………………. Weight ………………… Phone no …………………. Gestation age …………… Borg scale ……………. BMI ………………. Evaluation Sheet

Group A (RPT+ Insulin therapy)

Outcome variables:

1. Glucose level ………….
2. Delivery:

   i) Normal delivery ii) C-Section
3. APGAR Score:

   i) 1st min ……………. ii) 5th min …………….
4. Gestational age at birth ………

Outcome variables:

GROUP B (RPT+ Antenatal exercises+ Insulin therapy)

1. Glucose level ………….
2. Delivery:

   i) Normal delivery ii) C-Section
3. APGAR Score:

   i) 1st min ……………. ii) 5th min ……………. iii)
4. Gestational age at birth………

ELIGIBILITY:
Inclusion Criteria:

* Panel patients who are covered under medical facility provided by the company
* Booked cases
* Participant's Borg scale score 6 to 14
* Age 20-35 years
* 20-24 weeks of gestation
* Diagnosed case of GDM
* Primigravida
* BMI does not exceed 40 kg/m²

Exclusion Criteria:

* Females diagnosed with vascular complications (Preeclampsia, hemolysis etc.)
* Uncontrolled diabetes mellitus
* Autonomic dysfunction /Peripheral neuropathy (Damage to the nerves outside of the brain and spinal cord which effect sensations)
* Nephropathy or retinopathy (Damage to the small blood vessels of kidneys and eyes)
* Twins fetus
* Placenta Previa (placenta partially or totally covers the mother's cervix)
* Fetal anomalies
* Female choice for caesarean section
* Intrauterine growth retardation (fetal complication)
* Short cervix length
* Antepartum hemorrhage (bleeding from the genital tract)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Glucose level | 4 months
  Effect of antenatal exercise on glucose level was measured by test beta HbAc1 performed by gynecology department before delivery
mode of delivery | 4 months
  effect of antenatal exercise on type of delivery was studied as it was normal vaginal or caesarian section
APGAR Score | 4 months
  effect of antenatal exercise on APGAR score was studied which describe fetal health after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Anum Sattar, MPhil, Principal Investigator — student
Locations (1):
- Anumsattar8@Gmail.Com, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
all collected data will be share.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2021 data will available approximately
Access Criteria: Any one can access the data
URL: http://pubmed.gov